CLINICAL TRIAL: NCT06832722
Title: Multi-center, Randomized, Placebo-controlled, Double-blind Phase 1bTrial to Investigate Safety, Tolerability and Pharmacokinetics of Procizumab (PCZ; AK1967) in Patients With Cardiogenic Shock and Elevated Circulating Dipeptidyl Peptidase 3 (cDPP3) Concentrations
Brief Title: Procizumab (PCZ; AK1967) in Critical Cardiovascular Care
Acronym: PROCARD 1b
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 4TEEN4 Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-P1-002; 2024-518450-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-07; First posted 2025-02-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Shock, Cardiogenic
Keywords: Cardiogenic shock; Procizumab
MeSH Terms: conditions — Shock, Cardiogenic | interventions — procizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Procizumab (AK1967) 10mg/kg body weight (Active Comparator): 10 mg/kg body weight
  Interventions: Drug: AK1967 (Procizumab)
- Procizumab (AK1967) other dose regimen based on PK profile (Active Comparator): Other dose regimen based on PK profile
  Interventions: Drug: AK1967 (Procizumab)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK1967 (Procizumab) — DPP3 inhibition using the humanized monoclonal antibody AK1967 (Procizumab)
  Arms: Procizumab (AK1967) 10mg/kg body weight; Procizumab (AK1967) other dose regimen based on PK profile
Drug: Placebo — Application of placebo
  Arms: Placebo

SUMMARY:
The objective of this Phase 1b trial is to evaluate the safety and tolerability of procizumab, a monoclonal antibody under development for the treatment of cardiogenic shock (CS). CS is a life-threatening hypoperfusion of vital organs that frequently results in death. In addition to safety and tolerability, pharmacokinetics and pharmacodynamics of procizumab are evaluated to define the optimum phase 2 dose (P2D) of procizumab.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Diagnosis of CS due to ACS or CS of septic origin based on the following entry criteria:

  1. Need for ongoing vasopressors and/or to maintain a MAP ≥ 65 mmHg or SBP ≥ 90 mmHg
  2. Serum lactate ≥ 2.0 mmol/L
  3. Elevated DPP3 concentration

Exclusion Criteria:

* Patients who will be receiving vasopressors and/or inotropes for more than 16 hours prior to receiving the IMP.
* Patients below the age of 18 or above 75 years.
* Patients receiving Ang II and/or Levosimendan.
* Patients with known allergies or hypersensitivity to the IMP or its excipients (including known lactose hypersensitivity) or any related medication.
* Stroke or transient ischemic attack within the last 3 months.
* SCAI Stage E or most severe SCAI D including circulatory collapse refractory to treatment and/or loss of consciousness.
* Patients with SOFA score 12 and above in Part 1; SOFA score 14 and above in Part 2/3.
* Patients on MCS. MCS includes any type of mechanical support device including IAoBP, left ventricular assist device of any type or kind and renal replacement or mechanical support devices of any type or kind.
* Patients exceeding a maximum body weight of 120 kg.
* CPR lasting more than 15 minutes and the patient is not fully conscious at randomization.
* Primary hypertrophic or restrictive cardiomyopathy or systemic illness known to be associated with infiltrative heart disease.
* Shock triggered primarily by a correctable causality such as significant arrhythmia (inclusive of atrial fibrillation as the main reason for admission), severe anemia, pulmonary embolism, exacerbation of chronic obstructive pulmonary disease, or device implantation, or over-diuresis as a cause of hypotension.
* Pericardial constriction or active pericarditis.
* Patients suffering from CS due to myocarditis.
* Significant ventricular arrhythmia prior to screening (such as sustained ventricular tachycardia or ventricular fibrillation) or ICD shock within the past month or history of sudden death within the last 6 months.
* CRT, ICD, or pacemaker implantation within the past month.
* Sustained SBP > 120 mmHg during the hour prior to randomization.
* Cor pulmonale or other causes of isolated right-sided HF or not related to left ventricular dysfunction.
* Known severe renal disease before admission requiring dialysis or known eGFR prior to admission < 20 ml/min/1.73 m2.
* Laboratory exclusions:

  1. Hemoglobin < 8.5 g/dl
  2. Platelet count < 30,000/µl for CS from septic origin
  3. Platelet count < 100,000/µl for CS from ACS origin
  4. Serum potassium > 5.7 mmol/L or < 3.3 mmol/L
* Severe chronic pulmonary or thyroid disease.
* Patients with untreated sepsis.
* Patients with severe valvular heart diseases. This includes any moderate or severe stenotic valvular disease, any moderate or severe aortic or pulmonary regurgitation and severe mitral or tricuspid regurgitation.
* Patients experiencing hemorrhagic, hypovolemic, obstructive, anaphylactic shock or shock related to intoxication or any other reason for shock besides ischemic or septic/ inflammatory causes.
* Patients who have undergone chemotherapy within 30 days prior to trial entry.
* Patients receiving chronic corticosteroid treatment equivalent to a prednisone dose of 10 mg or higher per day, or an equivalent dose of another corticosteroid or any other anti-inflammatory or inflammation suppressing medications such as interleukin blockers, methotrexate or other such therapies.
* Patients who have undergone any form of surgery in the last 7 days will be excluded from the trial or analysis, except 1) minor surgeries such as cosmetic surgeries, skin surgery and dental surgery and 2) primary post operative peritonitis, which are allowed.
* Women who are pregnant or breastfeeding.
* Patients who are currently enrolled in another clinical trial, or who have participated in such trials within one month prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Reported number of treatment-emergent adverse events from start of Procizumab administration up until the last follow-up visit after Procizumab administration | 30 days

SECONDARY OUTCOMES:
Pharmacokinetics defined as plasma-time concentration of procizumab | 30 days
Pharmacodynamics defined as cDPP3 concentration | 30 days
Pharmcodynamics defined as cDPP3 activity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, Professor, Principal Investigator — Hôpital Lariboisière, Paris France
Locations (16):
- Belgium (2):
  - Heart Center Aalst, AZORG, Aalst
  - University Hospital Saint Pierre, Brussels
- Czechia (4):
  - University Hospital and Medical Faculty of Pilsen, Pilsen
  - Charles University Motol University Hospital, Prague
  - General University Hospital in Prague - FVN, Prague
  - Institute of Clinical and Experimental Medicine - IKEM, Prague
- France (5):
  - University Hospital Avicenne AP-HP, Bobigny
  - University Hospital Lille - Institut Cœur Poumon, Lille
  - University Hospital - Dupuytren Limoges, Limoges
  - Regional University Hospital Nancy - Hopitaux de Brabois, Nancy
  - Lariboisière Hospital AP-HP, Paris
- Radboud University Medical Center, Nijmegen, Netherlands
- Poland (4):
  - Uniersytecki Szpital Kliniczny w Białystoku, Bialystok
  - Górnośląskie Centrum Medyczne w Katowicach / Śląski Uniwersytet Medyczny w Katowicach, Katowice
  - Clinical University Hospital Poznań, Poznan
  - J. Mikulicz Radecki Clinical University Hospital Wrocław, Wroclaw

IPD SHARING:
Plan to Share IPD: No